CLINICAL TRIAL: NCT03069638
Title: Intranasal Dexmedetomidine Sedation During Intra-articular Joint Injections in Pediatric Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Outi Peltoniemi, PhD, Senior physician in Oulu University Hospital at the Department of Pediatrics (PICU), University of Oulu
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INDEXJIA
Record Dates: First submitted 2016-12-20; First posted 2017-03-03 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Juvenile Idiopathic Arthritis; Joint Inflammation
Keywords: sedation; pediatrics; intranasal sedation; dexmedetomidine; dinitrous oxide; intra-articular joint injection
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis | interventions — Dexmedetomidine; Tranquilizing Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal dexmedetomidine (Experimental): Dexmedetomidine is given once 4 micrograms per kilogram intranasally. If the sedation is not successful another 2 microgram per kilogram intranasal dose is given. Intravenous dexmedetomidine solution is administrated intranasally with MAD nasal drug delivery device and a syringe.
  Interventions: Drug: Dexmedetomidine; Drug: Sedatives/Hypnotics,Other
- Nitrous oxide inhalation (Active Comparator): Dinitrousoxide (N2O) is given with Livopan administrating device. Livopan consists of 50% oxygen and 50% nitrous oxide. Gas mixture is inhaled 5 minutes before the injection procedure and during the injection procedure.
  Interventions: Drug: Dexmedetomidine; Drug: Sedatives/Hypnotics,Other

INTERVENTIONS:
Drug: Dexmedetomidine — Intranasal administration of dexmedetomidine as a procedural sedation (intra-articular joint injection)
Drug: Sedatives/Hypnotics,Other — Inhaled dinitrous oxide as procedural sedation (intra-articular joint injection)
  Other Names: Dinitrous oxide

SUMMARY:
The main objective of this study is to evaluate the effectivity of intranasal dexmedetomidine sedation during intra-articular injection therapy. Intranasal dexmedetomidine is compared with dinitrous oxide (N2O) which has already been proven safe and effective sedation method during painful procedures in pediatric patients.

In earlier studies the median VAS during intra-articular corticosteroid injections with patients receiving nitrous oxide has been 3 (Uziel et al 2008). Study hypothesis is that with intranasal dexmedetomidine sedation the VAS pain levels will be 1 unit lower.

ELIGIBILITY:
Inclusion Criteria:

* Patient age between ages 1year to 18 years
* A joint inflammation in 1-5 joints needing intra-articular corticosteroid injection diagnosed by pediatric rheumatologist

Exclusion Criteria:

* Patients under the age of 1year and over the age of 18years are excluded as well as patients needing injection therapy to more than 5 joints.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Visual Analog scale (VAS) | The VAS score is assessed after procedure when the patients have recovered from the sedation and are being discharged. The time of discharge is 1 to 5 hours after the injection procedure.
  VAS scores of the pain experienced during the procedure are evaluated as a primary outcome.

SECONDARY OUTCOMES:
Blood pressure | Assessed in every 5 minutes 20 minutes before the drug administration and for six hours after the drug administration.
  Blood pressure is measured indirectly with a cuff
Heart rate | Assessed in every 5 minutes 20 minutes before the drug administration and for six hours after the drug administration.
  Heart rate is monitored by contiunously assessing Electro Cardiogram
Heart rate | Assessed in every 5 minutes 20 minutes before the drug administration and for six hours after the drug administration.
  Heart rate is monitored by contiunously assessing pulse oxymetry.
Respiratory rate | Assessed in every 5 minutes 20 minutes before the drug administration and for six hours after the drug administration.
  Respiratory rate is detected by capnometer or assessed manually
FLACC | Before the injection procedure, during the injection procedure, 5 and 10 minutes after the procedure and when the patient is being discharged.
  The Face, Legs, Activity, Cry, Consolability scale or FLACC scale is a measurement used to assess pain for children
COMFORT-B | Assessed 20 minutes before the drug administration and in every 15 minutes for six hours after the drug administration and during the injection procedure and 5 and 10 minutes after the injection.
  COMFORT-B is a sedation scale used to assess the level of sedation in children.
Capnometry | Assessed continuously 20 minutes before the drug administration and for six hours after the drug administration.
  Capnometry detects the exhaled carbon dioxide.
Pulse oxymetry | Oxygen saturation by pulse oxymetry is measured continuously 20 minutes before the drug administration and for six hours after the drug administration.
  Oxygen saturation is measured by pulse oxymetry
Visual Analog scale (VAS) | At the follow up visit which usually is 2-12 weeks after the injection.
  VAS scores of the pain experienced during the procedure evaluated at the follow up visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu university hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No